CLINICAL TRIAL: NCT05115994
Title: Antihypertensive and PAP Treatment in Obstructive Sleep Apnea Patients With Hypertension -Long Term Prospective Analysis on Cardiovascular Events or Death (AHPAP-MCE/Death)
Brief Title: Antihypertensive and PAP Treatment in Obstructive Sleep Apnea Patients With Hypertension (AHPAP)
Acronym: AHPAP
Status: Active, not recruiting | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Principal Investigator, Sven Svedmyr, Principal investigator, MD Sahlgrenska University Hospital, PhD student Gothenburg University, Specialist internal medicine, Vastra Gotaland Region
Other Study IDs: AHPAP-MCE/death
Record Dates: First submitted 2021-10-07; First posted 2021-11-10 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Obstructive Sleep Apnea; Hypertension; Death, Cardiac; Treatment Compliance; Heart Failure; Stroke
Keywords: Continous positive airway pressure; Antihypertensive treatment; Risc prevention
MeSH Terms: conditions — Sleep Apnea, Obstructive; Hypertension; Death; Patient Compliance; Heart Failure; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Hypertensive OSA patients, high PAP compliance: Hypertensive OSA patients using their PAP device for at least 4 hrs/night
  Interventions: Device: Continous positive airway pressure
- Hypertensive OSA patients, low PAP compliance: Hypertensive OSA patients using their PAP device for less than 4 hrs/night
  Interventions: Device: Continous positive airway pressure
- Intra oral device treatment: Hypertensive OSA patients treated with IOD
  Interventions: Device: Continous positive airway pressure
- Untreated OSA hypertensive patients: Hypertensive OSA patients not using PAP or IOD
- Hypertensive patients without OSA: Control population from QregPV without OSA

INTERVENTIONS:
Device: Continous positive airway pressure
  Other Names: Antihypertensive pharmacological treatment
  Groups: Hypertensive OSA patients, high PAP compliance; Hypertensive OSA patients, low PAP compliance; Intra oral device treatment

SUMMARY:
The investigators will perform a long term registry based prospective analysis on incidence of major cardiovascular events or death in hypertensive patients with obstructive sleep apnea .

Effects of PAP (positive airway pressure) compliance, antihypertensive medication and blood pressure control will be investigated in the study.

DETAILED DESCRIPTION:
By using swedish personal ID numbers the investigators can combine data from several quality registries in Sweden and will start with patients from a primary care registry (QregPV) that had or received a hypertension diagnosis during the period 2008-2012. The investigators will compare those who got an OSA diagnosis in the SESAR (Swedish sleep apnea registry) stratified by high/low PAP compliance with an intraoral device group, a non treated OSA group as well as a control group without OSA until 2021. Main outcome variables will be major cardiovascular events or death. Outcome data will be collected from the National Patient Registry and Cause of death registry.

Groups will be matched by propensity score for known confounders. Secondary analysis will consider modifying effect of different antihypertensive drugs (the Swedish Prescribed Drug Register, type of therapy; DDD comparison) and the actual degree of hypertension control (blood pressure levels) on CV risk. It is intended to stratify the analysis for BP levels in order to evaluate if lower BP targets further reduce CV risk in hypertensive OSA patients. These analyses will likely be reported in separate publications.

HYPOTHESIS

1. PAP treatment in hypertensive OSA patients reduces the long term risk of major cardiovascular events (MCE) and premature death. The risk reduction is modified by PAP compliance, hypertension control and OSA severity.
2. In hypertensive OSA patients, the investigators previously identified betablockade as a drug class leading to better pressure control (1). The investigators hypothesize that any risk reduction by PAP treated OSA is influenced by the types of antihypertensive drugs used.
3. Lower blood pressure targets (ie better BP control) may reduce the risk of cardiovascular events in PAP treated OSA patients.

ELIGIBILITY:
Inclusion Criteria:

* All hypertensive and obstructive sleep apnea patients present in QregPV and SESAR 2008-2021.

Exclusion Criteria:

* Patients in the hypertensive control group (without OSA) will be excluded if they have OSA diagnosis but are not present in the SESAR registry.
* Subjects with missing data on any of the variables in the fitted model unless the missing data can be accurately imputated.
* Patients with low life expectancy (Age>75 at study start, malignant disease).
* Patients no longer living in VGR 2021.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Propensity score matched registry cohorts
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2008-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Major cardiovascular event (MCE) or death | First incidence during study, ie within 156 months (13 yrs) maximum
  First incidence of new myocardial infarction, cardiac failure, stroke or death (cardiovascular and all)

SECONDARY OUTCOMES:
Blood pressure control | at study end (latest available BP measurements up to december 2021), ie within 156 months (13 yrs) maximum
  According to ESC/EHC 2018 guidelines
New incidence of atrial fibrillation | First incidence during study, ie within 156 months (13yrs) maximum
  New diagnosis from patient registry

OTHER OUTCOMES:
Subanalysis of MCE/death incidence, stratified by blood pressure levels | First incidence during study, ie within 156 months (13yrs) maximum
  Does baseline and end of study BP levels influence our outcomes? Does lower BP targets further reduce the outcome risc?

CONTACTS AND LOCATIONS:
Overall Officials: Sven Svedmyr, MD, Principal Investigator — Vastra Gotalands regionen, Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Västra Götaland County, Sweden

REFERENCES:
- [Background] Svedmyr S, Hedner J, Zou D, Parati G, Ryan S, Hein H, Pepin JL, Tkacova R, Marrone O, Schiza S, Basoglu OK, Grote L; European Sleep Apnea Database (ESADA) study group. Superior hypertension control with betablockade in the European Sleep Apnea Database. J Hypertens. 2021 Feb 1;39(2):292-301. doi: 10.1097/HJH.0000000000002629. PMID 33031170